CLINICAL TRIAL: NCT02992249
Title: Prospective Evaluation of the ReCell® Autologous Cell Harvesting Device For Specific Compassionate Use Cases
Status: Completed | Type: Observational
Sponsor: Avita Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CTP004
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective uncontrolled observational study to evaluate clinical outcomes following use of the ReCell Autologous Cell Harvesting Device (ReCell) as an adjunct for closure (re-epithelialization) as a treatment of life-threatening wounds requiring grafting for closure, and associated skin graft donor sites, in patients who lack adequate available skin to harvest for conventional grafting. Treatment with the ReCell device may be performed as part of a single operative procedure, or multiple staged procedures as deemed clinically necessary. Adverse events associated with the use of the ReCell device/cell suspension will be documented. Subjects will be followed for 1 year following ReCell treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient requires treatment of a life-threatening wound requiring grafting.
* Patient has inadequate available skin to harvest for conventional skin grafting.
* The treating investigator has determined 1) that there is no suitable alternative therapy that would be adequate to meet the patient's medical need; and 2) the risk associated with use of the ReCell device is no greater than the probable risk from the disease or condition.
* In the treating investigator's opinion and with consideration of the severity of the patient's health status, the patient has the potential to realize benefits from the application of the ReCell device.
* Patient is hemodynamically stable.
* The patient (or legal representative) is able to read and understand instructions and give informed consent.

Exclusion Criteria:

* The patient has active infection at the proposed ReCell treatment site.
* The patient is unable to follow the protocol.
* The patient has a known hypersensitivity to trypsin or Compound Sodium Lactate for Irrigation (Hartmann's) solution.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a prospective uncontrolled observational study to evaluate clinical outcomes following use of the ReCell Autologous Cell Harvesting Device (ReCell) as an adjunct for closure (re-epithelialization) as a treatment of life-threatening wounds requiring grafting for closure, and associated skin graft donor sites, in patients who lack adequate available skin to harvest for conventional grafting.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2019-05 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Wound Healing | Wound healing assessed at all study visits
  > 95% epithelialization with a contiguous layer of viable epithelium

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - University of South Alabama Department of Surgery, Mobile, Alabama
  - Arizona Burn Center at Maricopa Integrated Health Systems, Phoenix, Arizona
  - University of California San Diego Regional Burn Center, San Diego, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Grady Memorial Hospital, Atlanta, Georgia
  - Joseph M Still Research Foundation, Augusta, Georgia
  - Richard M. Fairbanks Burn Center at Eskenazi Health, Indianapolis, Indiana
  - Baton Rouge General Regional Burn Center, Baton Rouge, Louisiana
  - University Medical Center, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Walter Reed National Military Medical Center Bethesda, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Shriner's Boston, Boston, Massachusetts
  - MS Burn & Reconstruction Center, Merit Health Central, Jackson, Mississippi
  - University of Missouri Health Care, Columbia, Missouri
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Mercy General Burn Center - Springfield, Springfield, Missouri
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - U.S.Army Institute of Surgical Research, Fort Sam Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No